CLINICAL TRIAL: NCT06183476
Title: Circadian Amplification in Diabetic Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1387
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: Amplify-RHYTHM focuses on timed light exposure and weekly remote coaching session to optimize circadian and sleep behaviors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Amplify-RHYTHM will consist of two main components: 1) timed light exposure, 2) weekly remote coaching session.
  Interventions: Behavioral: Amplify-RHYTHM

INTERVENTIONS:
Behavioral: Amplify-RHYTHM — Amplify-RHYTHM will have two main components: 1) timed light exposure (increase light in the morning, blue light reduction in the evening and eye masks at night), 2) weekly remote coaching session by psychologist to optimize circadian and sleep behaviors

SUMMARY:
This study will test the effects of a 6-week comprehensive circadian optimization intervention Amplify-RHYTHM in patients with diabetic retinopathy. The outcomes of interest are objective and subjective sleep parameters, evening salivary cortisol and melatonin levels, and glucose parameters from continuous glucose monitoring

DETAILED DESCRIPTION:
This study will test the effects of a 6-week comprehensive circadian optimization intervention Amplify-RHYTHM in patients with diabetic retinopathy. The two main components of the intervention are timed light exposure and weekly remote coaching session by psychologist to optimize circadian and sleep behaviors. The outcomes of interest are objective and subjective sleep parameters, evening salivary cortisol and melatonin levels, and glucose parameters from continuous glucose monitoring

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* a history of at least moderate non-proliferative diabetic retinopathy
* would like to improve sleep
* own a smartphone compatible with fitbit.

Exclusion Criteria:

* Use of melatonin
* Use of antipsychotics
* Use of more than one antidepressant. The dose of which needs to be stable for 6 weeks.
* illicit drug use
* night shift work or travel beyond 2 time zones in the month before enrollment
* end stage renal disease requiring renal replacement therapy
* history of stroke or transient ischemic attacks
* history of dementia or memory impairment
* uncontrolled congestive heart failure or recent hospitalization for cardiac condition (6 months)
* chronic obstructive pulmonary disease requiring oxygen
* severe chronic liver disease such as cirrhosis
* ongoing treatment for major medical problems such as cancer
* history of severe hypoglycemia defined as hypoglycemic episodes requiring assistance from others within the past six months.
* Regular use of sedatives and hypnotics (>2 times/ month).
* clinically significant epiretinal membranes, clinically significant lens opacities, or cystoid macular edema, iris neovascularization, iris atrophy, or an asymmetrically shaped pupil, nuclear sclerotic, posterior subcapsular, or cortical lens opacities greater than 2+, a history of pan-retinal photocoagulation.
* Significant depressive symptoms as assessed by PHQ-8 questionnaire (score >14)
* No health insurance coverage
* History of untreated severe OSA.
* Uncontrolled hypertension (blood pressure ≥ 160/100 mmHg),
* Uncontrolled diabetes (A1C ≥ 11%)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Sleep | baseline and 6-week
  Objective and Subjective Sleep Parameters

SECONDARY OUTCOMES:
Salivary melatonin and cortisol | baseline and 6-week
  Evening salivary melatonin and cortisol
Glucose levels | baseline and 6-week
  Glucose from continuous glucose monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No